CLINICAL TRIAL: NCT04180878
Title: Promoting Appropriate Weight Gain Pregnant Women
Acronym: GRUVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13749
Record Dates: First submitted 2019-11-14; First posted 2019-11-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy
Keywords: Gestational weight gain; Physical activity
MeSH Terms: conditions — Gestational Weight Gain; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): Participants in this group were informed to continue to receive usual care.
- Intervention Arm (Experimental): Received an interactive physical activity monitoring system (the Gruve®).
  Interventions: Behavioral: Intervention
- Intervention Arm 2 (Experimental): Received an interactive physical activity monitoring system (the Gruve®) and group based phone counseling (GBPC).
  Interventions: Behavioral: Intervention 2

INTERVENTIONS:
Behavioral: Intervention — Participants received a interactive physical activity monitoring system that allowed study personnel to monitor their activity level.
  Arms: Intervention Arm
Behavioral: Intervention 2 — Participants received an interactive physical activity monitoring system, an electronic scale to report weekly body weight, weekly hour long conference calls with structured interactive educational lessons led by Health Educator, dietary recalls were completed at three different time points during their participation, and study personnel monitored physical activity levels weekly.
  Arms: Intervention Arm 2

SUMMARY:
The purpose of this study is to learn if engaging in group based phone counseling (GBPC) and an interactive physical activity monitoring system can help pregnant women gain an appropriate amount of weight during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 12-16 weeks pregnant
* Pre-pregnancy BMI between 22 kg/m2 to 45 kg/m2

Exclusion Criteria:

* Diabetes
* Pre-eclampsia
* Hypertension
* Other metabolic abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2016-02-03 (Actual)

PRIMARY OUTCOMES:
Excessive gestational weight gain | During Pregnancy - 18-36 week gestational age
  Proportion of excessive gestational weight gain based on weight gain guidelines.

SECONDARY OUTCOMES:
Gestational weight gain | During Pregnancy - 18-36 week gestational age
  Total weight change during pregnancy
Infant fat mass | 1-4 days after birth
  Infant fat mass

CONTACTS AND LOCATIONS:
Overall Officials: Holly R Hull, PhD, Principal Investigator — University of Kansas Medical Center